CLINICAL TRIAL: NCT00228982
Title: A Phase III, Randomized, Double-Blind Study of Ceftobiprole Versus Comparator in the Treatment of Complicated Skin and Skin Structure Infections
Brief Title: Ceftobiprole in the Treatment of Resistant Staphylococcus Aureus Skin and Skin Structure Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR005038; BAP00154 (Other: Basilea Pharmaceutica International Ltd.)
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Skin Diseases, Infectious; Skin Diseases, Bacterial; Staphylococcal Skin Infections
Keywords: Complicated Skin Infections; Infectious Skin Diseases; Bacterial Skin Diseases; Staphylococcal Skin Infections; Cephalosporin
MeSH Terms: conditions — Skin Diseases, Infectious; Skin Diseases, Bacterial; Staphylococcal Skin Infections | interventions — ceftobiprole medocaril; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftobiprole medocaril (Experimental): Ceftobiprole medocaril 500mg q12h as 1h infusion, 7-14d
  Interventions: Drug: Ceftobiprole medocaril
- Vancomycin (Active Comparator): Vancomycin 1g q12h as 1h infusion, 7-14d
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Ceftobiprole medocaril
  Arms: Ceftobiprole medocaril
Drug: Vancomycin
  Arms: Vancomycin

SUMMARY:
The purpose of this study is to compare the clinical cure rate of ceftobiprole medocaril versus a comparator in the treatment of patients with complicated skin and skin structure infections.

DETAILED DESCRIPTION:
Ceftobiprole medocaril is a cephalosporin antibiotic with anti-MRSA (Methicillin-Resistant Staphylococcus Aureus) activity. Ceftobiprole medocaril is not yet approved for the treatment of complicated skin and skin structure infections. This is a randomized, double-blind, multicenter study of ceftobiprole medocaril plus placebo versus a comparator to assess the effectiveness and safety of ceftobiprole medocaril in patients with complicated skin and skin structure infections. The patients will be randomized to ceftobiprole medocaril plus placebo or a comparator. The primary endpoint is the clinical cure rate of ceftobiprole medocaril at the test-of-cure visit. The patients will receive either ceftobiprole medocaril plus placebo or a comparator for 7 to 14 days (unless extended at discretion of medical monitor).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an infection consistent with complicated skin and skin structure infections.

Exclusion Criteria:

* Known or suspected hypersensitivity to any study medication
* Any known or suspected condition or concurrent treatment contraindicated by the prescribing information
* Previous enrollment in this study
* Treatment with any investigational drug within 30 days before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 784 (Actual)
Dates: Start 2004-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Clinical outcome (cure, failure, not evaluable) at 7-14 days after the end of therapy. | 7 weeks

SECONDARY OUTCOMES:
Microbiological outcome at 7-14 days after the end of therapy. Clinical and microbiological outcome at late follow-up visit. Evolution of signs and symptoms of disease. Time to clinical cure. Safety and tolerability evaluations during the study. | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.